CLINICAL TRIAL: NCT03462667
Title: Intensive Preoperative Ostomy Education for the Radical Cystectomy Patient
Acronym: StomABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00142039
Record Dates: First submitted 2018-02-23; First posted 2018-03-12 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Stoma Ileostomy
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stoma Boot Camp (Experimental): Participants will attend the Stoma Boot Camp session prior to surgery.
  Interventions: Behavioral: Stoma Boot Camp
- Regular Care (Active Comparator): Participants will receive normal standard of care prior to surgery.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Stoma Boot Camp — Educational session designed to prepare people for living life with a stoma.
  Arms: Stoma Boot Camp
Other: Standard of Care — Patients receive normal pre-surgery standard of care.
  Arms: Regular Care

SUMMARY:
The purpose of this study is to learn if the stoma boot camp is a good and effective way to help people adapt to life with a stoma after surgery.

DETAILED DESCRIPTION:
Bladder cancer is the fifth most common cancer in the USA. The primary treatment for invasive bladder cancer is a radical cystectomy (RC) with a urinary diversion. Patients that have this procedure must deal with a stoma that requires daily care and manual skills. A stoma is an artificial opening that allows urine to pass from the ureters outside the body. Having a surgery that results in a stoma can dramatically change a person's life.

This study is being done to test a new education session called the stoma boot camp. The session was created to help people deal with changes in their post-surgery life and living with a stoma.

The session requires a one time visit to the study site and lasts about two hours. Participants can bring a support person to the boot camp if they choose. During the two hour session, nurses will provide teaching, counseling, and hands on practice with an artificial stoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be presumed to undergo a radical cystectomy with ileal conduit diversion
* Diagnosis of bladder cancer

Exclusion Criteria:

* Patients undergoing a radical cystectomy with ileal conduit for any reason other than bladder cancer will not be allowed to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Ostomy adjustment scale | Change from Baseline to 30 Days After Date of Surgery
  The Ostomy Adjustment Scale evaluates a person with an ostomy following surgery. The instrument consists of 34 statements. Scores range from a minimum of 34 to a maximum of 204. The higher the score, the better the person's perceived adjustment.

SECONDARY OUTCOMES:
Length of hospital stay | Date of Admission to Date of Discharge, up to 7 days
  Measured as the date of admission to discharge.
Count of un-planned stoma-related interventions in community after discharge | 30 Days After Date of Surgery
  Unplanned stoma-related interventions will include any admission to any hospital after being discharged, from the time the patient goes home up until 30 days after the date of the surgery, along with any stoma related visit outside of the normal follow-up pathway to a clinic or any stoma related phone calls received by urology or ostomy staff.

CONTACTS AND LOCATIONS:
Overall Officials: Moben Mirza, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States